CLINICAL TRIAL: NCT01268267
Title: Clinical Trial Protocol for Ninja 2 System With TATSU Sensor
Brief Title: Performance of an Investigational Blood Glucose Monitoring System in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2010-008-01
Record Dates: First submitted 2010-12-28; First posted 2010-12-30 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the System (Experimental): Untrained subjects with diabetes obtained capillary fingerstick, palm, and forearm blood and performed Blood Glucose (BG) tests using an investigational blood glucose monitoring system (development name Ninja 2).
  Interventions: Device: Ninja 2 Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: Ninja 2 Investigational Blood Glucose Monitoring System — Untrained subjects with diabetes performed Blood Glucose(BG) tests from the subject's capillary blood obtained from fingerstick, palm, and forearm using the Ninja 2 investigational meter and an investigational sensor. All BG results were compared to a reference laboratory glucose method. Subjects' success at performing basic tasks using only the User Guide were rated by study staff.

SUMMARY:
The purpose of this study is to evaluate the performance and acceptability of an investigational blood glucose monitoring system, which includes meter and sensor strip.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and above
* Type 1 or type 2 diabetes
* Currently self-testing blood glucose at home at least twice daily
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Currently Pregnant
* Hemophilia or any other bleeding disorder
* Employee of competitive medical device company
* Cognitive disorder or other condition which, in the opinion of the investigator, would put the person at risk or seriously compromise the integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (1):
- AMCR Institute, Escondido, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the System: Untrained subjects with diabetes use an investigational blood glucose monitoring system.
Period: Overall Study
Arm/Group | Intended Users of the System
Started | 94
Completed | 93
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Intended Users of the System: Untrained subjects with diabetes use an investigational blood glucose monitoring system.One subject was found not to meet inclusion/exclusion criteria so subject was withdrawn and no data from this subject was evaluated.
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 93
Age, Customized [Mean (Full Range); unit: years] | 38.3 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 93

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Fingerstick Blood Glucose (BG) Results Within +/- 5 to 20mg/dL (<75 mg/dL) or Within +/- 5% to 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes tested subject fingerstick blood using an investigational blood glucose monitoring system (BGMS), which included an investigational meter and sensor. BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 5 to 20 mg/dL (for reference BG results <75mg/dL) or +/- 5 to 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 2 hours
Population: One subject was withdrawn from the study. One subject YSI reference sample was misidentified. Two subjects were not in steady state, required for the study. Four subjects' blood test data were thus not evaluable. The remaining 90 subjects tested 2 test strip lots on the BGMsystem. 2x90(180) test results were available.
Measure: Number; unit: Number of BG test results
Units Other Than Participants: Blood glucose test results
Groups:
- Intended Users of the System: Untrained subjects with diabetes use an investigational blood glucose monitoring system.One subject was found not to meet inclusion/exclusion criteria so subject was withdrawn and no data from this subject were evaluated.
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 90
Number analyzed (Blood glucose test results) | 180
Number of BG test results
  # within +/-15mg/dL(<75mg/dL) or 20% (>=75mg/dL) | 180
  # within +/-15mg/dL(<75mg/dL) or 15% (>=75mg/dL) | 179
  # within +/-10mg/dL(<75mg/dL) or 10% (>=75mg/dL) | 172
  # within +/-5mg/dL(<75mg/dL) or 5% (>=75mg/dL) | 138

2. Secondary Outcome: Numbers of Palm Blood Glucose (BG) Results Within +/- 5 to 20 mg/dL (<75 mg/dL) or Within +/- 5% to 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes used an investigational blood glucose monitoring system (BGMS) with subject capillary blood obtained from the palm. BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 5 to 20 mg/dL (for reference BG results <75mg/dL) or +/- 5% to 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 2 hours
Population: Five subjects were hypoglycemic (low blood glucose value). Since alternate-site palm testing by these subjects was not allowed in the study, palm data from these five subjects were not obtained/ not evaluable. The remaining 85 subjects tested 2 test strip lots on the BGM system. 2x85(170)test results were available.
Measure: Number; unit: Number of BG test results
Units Other Than Participants: BG test results
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 85
Number analyzed (BG test results) | 170
Number of BG test results
  # within +/-15mg/dL(<75mg/dL) or 20% (>=75mg/dL) | 166
  # within +/-15mg/dL(<75mg/dL) or 15% (>=75mg/dL) | 161
  # within +/-10mg/dL(<75mg/dL) or 10% (>=75mg/dL) | 143
  # within +/-5mg/dL(<75mg/dL) or 5% (>=75mg/dL) | 82

3. Secondary Outcome: Number of Subjects Rated as<=3 Performing Basic Meter Tasks (Labeling Comprehension)
Description: Subjects reviewed the instructions for use (User Guide and Quick Reference Guide) to learn to use the system. Study staff then observed and rated the subjects (1 to 4) on their success at performing the tasks. Scale: 1.Success in performing tasks correctly without assistance. 2.Successful with additional review of User Guide. 3.Successful with additional review and study staff assist similar to review of a specific function during a Customer Service call. 4.Subject did not perform task correctly and study staff intervention was required.
Time Frame: 2 hours
Population: For alternate-site palm and forearm testing tasks, 3 subjects with nonevaluable blood glucose data were not included. Only 90 participants were rated for those particular tasks.
Measure: Number; unit: participants
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 93
participants
  Turn meter on/off | 93
  Date and time set on meter | 93
  Normal control testing | 93
  Subject blood testing - fingerstick | 93
  Subject blood testing - palm (of 90) | 90
  Subject blood testing - forearm (of 90) | 90
  Understand underfill / ability to apply more blood | 93

4. Secondary Outcome: Numbers of Forearm Blood Glucose (BG) Results Within +/- 5 to 20 mg/dL (<75 mg/dL) or Within +/- 5% to 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes used an investigational blood glucose monitoring system (BGMS) with subject capillary blood obtained from the forearm. BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 5 to 20 mg/dL (for reference BG results <75mg/dL) or +/- 5% to 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 2 hours
Population: Since forearm testing by 5 hypoglycemic subjects (low blood glucose) was not allowed per the protocol, forearm data were not obtained/not evaluable for these subjects. Of the remaining 85 subjects, 83 tested 2 test strip lots(83x2) and 2 subjects tested 1 strip lot(2x1). A total of 168(166+2)test results were available.
Measure: Number; unit: Number of BG test results
Units Other Than Participants: BG test results
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 85
Number analyzed (BG test results) | 168
Number of BG test results
  # within +/-15mg/dL(<75mg/dL) or 20% (>=75mg/dL) | 158
  # within +/-15mg/dL(<75mg/dL) or 15% (>=75mg/dL) | 145
  # within +/-10mg/dL(<75mg/dL) or 10% (>=75mg/dL) | 125
  # within +/-5mg/dL(<75mg/dL) or 5% (>=75mg/dL) | 74

ADVERSE EVENTS:
Time Frame: Each subject participated for approximately 2 hours.
Arm/Group | Intended Users of the System
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 7/94
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the System (N=94)
hypoglycemia (Endocrine disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days